CLINICAL TRIAL: NCT07173374
Title: Stereotactic Centralized Ablative Radiotherapy for Locally Advanced Pancreatic Cancer: A Single-Arm Phase I Safety and Feasibility Study
Acronym: SCART-P
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Department Radiation Oncology, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-283-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Cancer
Keywords: SCART; Radiotherapy; Dose Escalation; Phase I Trial
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, phase I dose-escalation study using a standard 3+3 design to evaluate the safety and feasibility of SCART (Stereotactic Centralized Ablative Radiation Therapy) in patients with locally advanced pancreatic cancer.
Masking Description: This is an open-label, single-arm dose-escalation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCART Dose Escalation Arm (Experimental): Patients will receive SCART with escalating dose cohorts (10 Gy, 13 Gy, 16 Gy, and 19 Gy per fraction within the SCART region).
  Interventions: Radiation: SCART Dose Escalation Arm

INTERVENTIONS:
Radiation: SCART Dose Escalation Arm — Patients will receive SCART with escalating dose cohorts (10 Gy, 13 Gy, 16 Gy, and 19 Gy per fraction within the SCART region) using a standard 3+3 design. All patients will also receive background SBRT (25 Gy in 5 fractions) to the gross tumor volume and margin.

SUMMARY:
This is a single-arm, phase I clinical study designed to evaluate the safety and feasibility of SCART (Stereotactic Centralized Ablative Radiation Therapy) dose escalation in patients with locally advanced pancreatic cancer. Pancreatic cancer carries a dismal prognosis, and the majority of patients are not surgical candidates at diagnosis. Radiotherapy is an important local treatment modality, but conventional approaches have shown limited efficacy. SCART is intended to deliver higher ablative doses to the tumor core while minimizing toxicity to surrounding normal tissues. In this trial, eligible patients will receive SCART with escalating dose levels using a standard 3+3 design. The primary endpoints are to determine the dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD). Secondary endpoints include overall survival (OS), local control rate (LCR), and objective response rate (ORR).

DETAILED DESCRIPTION:
Pancreatic cancer is among the most aggressive malignancies and is associated with poor prognosis. The 5-year survival rate remains below 10%, and most patients present with unresectable disease at diagnosis. Radiotherapy plays a pivotal role in local disease control, yet conventional fractionated radiotherapy (CFRT) has demonstrated limited survival benefits. Stereotactic body radiotherapy (SBRT) allows delivery of higher biologically effective doses with improved local control, but further dose escalation is restricted by normal tissue tolerance.

SCART (Stereotactic Centralized Ablative Radiation Therapy) is an innovative technique that delivers ablative radiation doses to selected intratumoral sub-volumes while maintaining lower doses at the tumor periphery. This spatial dose distribution has the potential to induce bystander effects and enhance biological efficacy beyond that achievable with uniform SBRT.

This phase I study is designed to evaluate the safety and feasibility of SCART dose escalation in patients with locally advanced pancreatic cancer. Patients will be enrolled into sequential dose cohorts (10 Gy, 13 Gy, 16 Gy, and 19 Gy per fraction within the SCART region) using a standard 3+3 dose-escalation design. All patients will also receive background SBRT (25 Gy in 5 fractions) covering the gross tumor volume and margin.

The primary objective is to determine dose-limiting toxicities (DLTs) and establish the maximum tolerated dose (MTD) of SCART. Secondary objectives include overall survival (OS), local control rate (LCR), objective response rate (ORR), and treatment-related adverse events (AEs). Exploratory analyses will investigate potential biomarkers and immune response modulation associated with SCART.

The estimated enrollment is 12-24 patients, with an accrual period of 24 months and a minimum follow-up of 12 months.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-70 years, male or female. Histologically or cytologically confirmed diagnosis of pancreatic cancer. Locally advanced, unresectable disease without evidence of distant metastasis (based on imaging such as CT/MRI/PET-CT).

Eastern Cooperative Oncology Group (ECOG) performance status 0-1. Adequate bone marrow, liver, and renal function (per laboratory criteria). Life expectancy ≥ 3 months. Signed written informed consent prior to participation.

Exclusion Criteria:

- Evidence of distant metastasis. Prior abdominal radiotherapy. Prior systemic chemotherapy or immunotherapy within 4 weeks before enrollment. Concurrent participation in another interventional clinical trial. Severe comorbidities (e.g., uncontrolled cardiovascular, pulmonary, or infectious diseases).

Pregnant or breastfeeding women. Known history of other malignancies within the past 5 years (except adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ).

Any condition that, in the investigator's judgment, would interfere with patient safety or compliance with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within 90 days after completion of radiotherapy
  The maximum tolerated dose (MTD) of SCART (Stereotactic Centralized Ablative Radiation Therapy) will be determined using a standard 3+3 dose-escalation design. MTD is defined as the highest dose level at which the incidence of dose-limiting toxicities (DLTs), graded according to CTCAE v5.0, does not exceed 33% of patients in that cohort.
Dose-Limiting Toxicities (DLTs) | Within 90 days after completion of radiotherapy
  Incidence of dose-limiting toxicities (DLTs) graded according to the National Cancer Institute Common Terminology CTCAE v5.0. DLTs will be evaluated during the dose-escalation phase to assess the safety of SCART (Stereotactic Centralized Ablative Radiation Therapy).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 12 months after enrollment
  Overall survival will be defined as the time from the start of SCART treatment to death from any cause. Patients still alive at the time of analysis will be censored at the date of last follow-up.
Local Control Rate (LCR) | Up to 12 months after enrollment
  Local tumor control will be assessed according to RECIST v1.1 criteria based on radiographic imaging (CT/MRI). Local control rate will be calculated as the proportion of patients without local progression.
Objective Response Rate (ORR) | Up to 12 months after enrollment
  Objective tumor response will be evaluated using RECIST v1.1 criteria by imaging assessment.
Adverse Events (AEs) | Up to 12 months after enrollment
  Incidence and severity of treatment-related adverse events (AEs) will be graded according to CTCAE v5.0 during and after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song CW, Kim MS, Cho LC, Dusenbery K, Sperduto PW. Radiobiological basis of SBRT and SRS. Int J Clin Oncol. 2014 Aug;19(4):570-8. doi: 10.1007/s10147-014-0717-z. Epub 2014 Jul 5. PMID 24993673
- [Background] Gkika E, Firat E, Adebahr S, Graf E, Popp I, Radicioni G, Lo SS, Nestle U, Nicolay NH, Niedermann G, Duda DG, Grosu AL. Systemic immune modulation by stereotactic radiotherapy in early-stage lung cancer. NPJ Precis Oncol. 2023 Mar 2;7(1):24. doi: 10.1038/s41698-023-00358-z. PMID 36864234
- [Background] Timmerman RD, Herman J, Cho LC. Emergence of stereotactic body radiation therapy and its impact on current and future clinical practice. J Clin Oncol. 2014 Sep 10;32(26):2847-54. doi: 10.1200/JCO.2014.55.4675. Epub 2014 Aug 11. PMID 25113761
- [Background] Bouchart C, Navez J, Closset J, Hendlisz A, Van Gestel D, Moretti L, Van Laethem JL. Novel strategies using modern radiotherapy to improve pancreatic cancer outcomes: toward a new standard? Ther Adv Med Oncol. 2020 Jul 7;12:1758835920936093. doi: 10.1177/1758835920936093. eCollection 2020. PMID 32684987
- [Background] Lawlor RT, Mattiolo P, Mafficini A, Hong SM, Piredda ML, Taormina SV, Malleo G, Marchegiani G, Pea A, Salvia R, Kryklyva V, Shin JI, Brosens LA, Milella M, Scarpa A, Luchini C. Tumor Mutational Burden as a Potential Biomarker for Immunotherapy in Pancreatic Cancer: Systematic Review and Still-Open Questions. Cancers (Basel). 2021 Jun 22;13(13):3119. doi: 10.3390/cancers13133119. PMID 34206554
- [Background] Abravan A, Faivre-Finn C, Kennedy J, McWilliam A, van Herk M. Radiotherapy-Related Lymphopenia Affects Overall Survival in Patients With Lung Cancer. J Thorac Oncol. 2020 Oct;15(10):1624-1635. doi: 10.1016/j.jtho.2020.06.008. Epub 2020 Jun 14. PMID 32553694
- [Background] Treatment of locally unresectable carcinoma of the pancreas: comparison of combined-modality therapy (chemotherapy plus radiotherapy) to chemotherapy alone. Gastrointestinal Tumor Study Group. J Natl Cancer Inst. 1988 Jul 20;80(10):751-5. PMID 2898536
- [Background] Sultana A, Tudur Smith C, Cunningham D, Starling N, Tait D, Neoptolemos JP, Ghaneh P. Systematic review, including meta-analyses, on the management of locally advanced pancreatic cancer using radiation/combined modality therapy. Br J Cancer. 2007 Apr 23;96(8):1183-90. doi: 10.1038/sj.bjc.6603719. Epub 2007 Apr 3. PMID 17406358
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Chauffert B, Mornex F, Bonnetain F, Rougier P, Mariette C, Bouche O, Bosset JF, Aparicio T, Mineur L, Azzedine A, Hammel P, Butel J, Stremsdoerfer N, Maingon P, Bedenne L. Phase III trial comparing intensive induction chemoradiotherapy (60 Gy, infusional 5-FU and intermittent cisplatin) followed by maintenance gemcitabine with gemcitabine alone for locally advanced unresectable pancreatic cancer. Definitive results of the 2000-01 FFCD/SFRO study. Ann Oncol. 2008 Sep;19(9):1592-9. doi: 10.1093/annonc/mdn281. Epub 2008 May 7. PMID 18467316
- [Background] Loehrer PJ Sr, Feng Y, Cardenes H, Wagner L, Brell JM, Cella D, Flynn P, Ramanathan RK, Crane CH, Alberts SR, Benson AB 3rd. Gemcitabine alone versus gemcitabine plus radiotherapy in patients with locally advanced pancreatic cancer: an Eastern Cooperative Oncology Group trial. J Clin Oncol. 2011 Nov 1;29(31):4105-12. doi: 10.1200/JCO.2011.34.8904. Epub 2011 Oct 3. PMID 21969502
- [Background] Auclin E, Marthey L, Abdallah R, Mas L, Francois E, Saint A, Cunha AS, Vienot A, Lecomte T, Hautefeuille V, de La Fouchardiere C, Sarabi M, Ksontini F, Forestier J, Coriat R, Fabiano E, Leroy F, Williet N, Bachet JB, Tougeron D, Taieb J. Role of FOLFIRINOX and chemoradiotherapy in locally advanced and borderline resectable pancreatic adenocarcinoma: update of the AGEO cohort. Br J Cancer. 2021 Jun;124(12):1941-1948. doi: 10.1038/s41416-021-01341-w. Epub 2021 Mar 26. PMID 33772154
- [Background] Badiyan SN, Molitoris JK, Chuong MD, Regine WF, Kaiser A. The Role of Radiation Therapy for Pancreatic Cancer in the Adjuvant and Neoadjuvant Settings. Surg Oncol Clin N Am. 2017 Jul;26(3):431-453. doi: 10.1016/j.soc.2017.01.012. Epub 2017 May 11. PMID 28576181
- [Background] Fukumura D, Jain RK. Tumor microvasculature and microenvironment: targets for anti-angiogenesis and normalization. Microvasc Res. 2007 Sep-Nov;74(2-3):72-84. doi: 10.1016/j.mvr.2007.05.003. Epub 2007 May 18. PMID 17560615
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Strohl MP, Raigani S, Ammori JB, Hardacre JM, Kim JA. Surgery for Localized Pancreatic Cancer: The Trend Is Not Improving. Pancreas. 2016 May-Jun;45(5):687-93. doi: 10.1097/MPA.0000000000000511. PMID 26491905
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Klein AP. Pancreatic cancer epidemiology: understanding the role of lifestyle and inherited risk factors. Nat Rev Gastroenterol Hepatol. 2021 Jul;18(7):493-502. doi: 10.1038/s41575-021-00457-x. Epub 2021 May 17. PMID 34002083